CLINICAL TRIAL: NCT05769517
Title: PREDICTION OF GERMLINE BRCA 1/2 GENES PATHOGENETIC VARIANTS FROM HEALTHY OVARIES ULTRASOUND IMAGES: RADIOGENOMICS AS AN INNOVATIVE TOOL TO PREVENT BRCA-RELATED CANCERS
Brief Title: PREDICTION OF GERMLINE BRCA 1/2 GENES FROM HEALTHY OVARIES
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5505
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: BRCA Mutation; Ovarian Cancer; Ultrasound Therapy; Complications
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Germinal BRCA — We will conduct a multicenter prospective observational study aimed at automatically implementing the predictive model and collecting US images of healthy ovaries from patients tested for germline BRCA pathogenetic variants according to current indications.

SUMMARY:
The project aims at enhancing performance metrics and prospectively validating a radiogenomics model based on ovarian US images for predicting germline breast cancer susceptibility gene 1 and/or 2 (BRCA) status in women with healthy ovaries. The project is divided in two operational phases:

Retrospective phase

AIM 1: To define and implement a proper and fine-tuned image preprocessing pipeline on the existing dataset; AIM 2: To enlarge dataset size with new real images from different centers and apply data augmentation techniques, deep neural network models combined with the aforementioned handcrafted imaging features from radiomics analysis;

Prospective phase

AIM 3: To further cross-validate the predictive model on US images acquired prospectively in an observational multicenter study.

ELIGIBILITY:
Inclusion Criteria:

Availability of gBRCA1/2 test results

Transvaginal pelvic US performed providing at least one picture of one healthy ovary

US images stored in .dicom format.

Exclusion Criteria:

Personal diagnosis of OC

Ovarian abnormal findings (eg. ovarian endometriomas, dermoid cyst, ovarian cystoadenofibroma, ovarian borderline tumour…) with the exception of functional cysts at pelvic US

gBRCA1/2 testing results nor provided by an ISO 1589 accredited laboratory

Refusal to provide written informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: We will conduct a retrospective multicenter observational study aimed at collecting US images of healthy ovaries with known BRCA status.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Radiogenomics model for predicting germline breast cancer. | 36 months
  The project aims at enhancing performance metrics and prospectively validating a radiogenomics model based on ovarian US images for predicting germline breast cancer susceptibility gene 1 and/or 2 (BRCA) status in women with healthy ovaries.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No